CLINICAL TRIAL: NCT06829875
Title: Are We Providing Timely Access to Musculoskeletal Outpatient Therapy Services? an Exploratory Study
Acronym: MSk EATS
Status: Recruiting | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: 8851
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal
Keywords: access; waiting times; impact of wait; musculoskeletal pain; msk pain; musculoskeletal conditions; physiotherapy outpatients; podiatry outpatients; occupational therapy outpatients; musculoskeletal therapy services
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- service users entering waiting lists for outpatient musculoskeletal physiotherapy, podiatry and OY
  Interventions: Procedure: wait for outpatient appointment

INTERVENTIONS:
Procedure: wait for outpatient appointment — this is an observational study measuring impact of pain and function at start and end of wait for those waiting for care from outpatient physiotherapy occupations therapy and podiatry

SUMMARY:
Waiting times for NHS services are of growing public interest. This is because accessing some services is getting more difficult, and we know that longer waits can result in negative impacts for those waiting.

People in Wales waiting for care for their musculoskeletal problems are deemed to be cared for in good time if they get an appointment in less than 14 weeks. This target has been set by Welsh Government, for everyone who waits, no matter what condition they are waiting with and how that condition is affecting them.

We know that impact of wait for people with MSK problems can vary, from complete recovery, to worsening of their pain and function. The impact experienced seems to be influenced by factors such as their age and their mental health statusz\. This suggests that setting one target for all may not be the right thing to do. However, we don't yet know whether waiting over 14 weeks has a big effect on impact. We also don't know about the lived experience of those waiting, while they wait, despite knowing that learning this is vital to informing change.

We plan to study the impact of waiting for these services by asking those waiting to complete a survey that measures the impact of their msk problem, at the start and end of their wait, and then understanding how the scores correlate with length of time waited. We will also ask some of these people to document their experience as they wait. We hope that this will provide an understanding of how effective the current target is at measuring access to these services, and whether we need to think differently. People will be able to complete this work in their own home.

DETAILED DESCRIPTION:
Access to NHS and social care services has been of increasing public interest for many years. Increasing waits to services has been long documented, and the COVID-19 pandemic saw waiting times soar to an all time high. This is not favourable because of the known negative impacts experienced by the waiter, when waiting longer for the services they need. Improving access to services is not only a National Driver featured throughout policy (A Healthier Wales, 2018) but a legal obligation (Duty of Quality, 2023). Access to services in Wales has been studied by Welsh Government for decades. This is usually measured by the time taken in weeks from referral to treatment, and is supported to be necessary in some areas, whereby increased waiting time can result in morbidity, or mortality, for example, heart attacks and strokes.

Literature exploring impact with wait is lacking when considering many areas of health, for example musculoskeletal conditions. However, such services are also duty bound to report their waiting times to Welsh Government.

Outpatient MSk Therapy Services, for example, report how long each person waits before an initial appointment is offered, in number of weeks. An appointment offered within 14 weeks of referral is considered 'timely' and people waiting over this time are considered to be 'breaching'. How this target became to be considered significant is not publicly justified. The impact of those waiting over 14 weeks on the person waiting, is not known.

Impact exploring those waiting for treatment for musuculoskeletal disorders is extremely limited. However, preliminary, retrospective study during COVID-19 suggests that those waiting for these services during this time, experienced a diversity of impact, from symptom recovery to deterioration of condition. The variables observed differed between individuals, as opposing to differing lengths of wait, and seemed to be influenced by personal factors such as socioeconomic and mental health status. This provides an insight that impact of wait is variable between individuals and does not align with current study of accessibility subjecting all people to the same arbitrary target without knowing what happens around this time. We know that future health and social care services need to be sustainable for the NHS to survive. We know that we need to look at things differently, considering the quality of the care that is provided rather than the quantity, and we are duty bound to explore how the NHS is doing with respect to quality, using both qualitative and quantitative information, involving all stakeholders. We know that this is vital to inform positive system change. However, there is no current exploration into the experience of waiting for MSk services, in the eyes of the waiter, as they wait.

Understanding this may help us to understand what a future model of MSk Outpatient healthcare should look like with respect to accessibility, and implement a sustainable solution for future generations. This is assuming that our current understanding of wait is inadequate, or not appropriate, based on the information available communicating accessibility through use of an arbitrary, unjustified blanket target for all, which remains an unknown.

This research project aims to understand the impact of chronological wait for people waiting for Musculoskeletal Therapy Outpatient Services, with reference given to under and over 14 weeks, to understand if the current target is effective at communicating how we are doing in this domain. It will also explore the lived experience of waiting in the eyes of the waiter, and seeks to understand whether this understanding aligns with what we see when studying impact of wait chronologically, with a view to provide a quality rich understanding of the impact of waiting for these services, and provide a direction of travel for future study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over
* have entered a waiting list for outpatient podiatry, occupational therapy or physiotherapy with a musculoskeletal complaint
* able to provide informed consent
* be able to read and write english

Exclusion Criteria:

* are considered a vulnerable adult
* exhibit additional communication needs, to include but not limited to, language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people residing in the remit of Cardiff and Vale University Health Board, entering the waiting list of Outpatient Musculoskeletal Physiotherapy, Occupational therapy or Podiatry
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
musculoskeletal Health Questionnaire | from enrolment until the end of wait - currently up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara P James, MSc, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Cardiff and Vale University Healthboard, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No
CI handling all participant information. Feasibility study